CLINICAL TRIAL: NCT01268085
Title: Radiation Safety Alert- A Randomized Controlled Trial
Brief Title: Radiation Safety Alert
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Error in randomization resulted in early study termination.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10-10-330
Record Dates: First submitted 2010-12-15; First posted 2010-12-29 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Radiation Safety
Keywords: Radiation Safety; Computerized Physician Order Entry; Decision Support; Cat Scans

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation Safety Alert (Experimental): A provider placing an electronic order for a CAT scan will receive a radiation safety pop-up alert with a message about the dangers of cumulative ionizing radiation, the patient's cumulative CAT scan history, and the most recent imaging test from any modality of the same body part.
  Interventions: Other: Radiation Alert
- Control (Active Comparator): Parallel control with no intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: Radiation Alert — A radiation safety pop-up alert with a message about the dangers of cumulative ionizing radiation, the patient's cumulative CAT scan history, and the most recent imaging test from any modality of the same body part
  Arms: Radiation Safety Alert
Other: Control — Control with no inverention
  Arms: Control

SUMMARY:
In recent years, multiple articles have highlighted the increased risk of developing cancer from ionizing radiation. The risk increases with higher radiation doses, and accumulates with repeated scans.

Hospitals with computerized physician order entry systems (CPOE) have the unique opportunity to use decision support on radiation safety to influence a physician's ordering practice in real-time. An ideal decision support tool for radiation safety will educate the physician about the dangers of cumulative ionizing radiation, present the patient's image history, and guide the provider to the best modality that meets the patient's diagnostic needs with as little radiation exposure as possible. The design challenge is to create a decision support tool that appropriately protects the investigators patients from overutilization of CAT scans, without inadvertently leading to underutilization of CAT scans or inappropriate utilization of alternative tests.

This research protocol proposes to study one such design at a large, academic medical center.

DETAILED DESCRIPTION:
Ever since the 1979 Nobel Prize was awarded to Cormack and Hounsfield for the development of computer assisted tomography (CAT scans, this technology has revolutionized the practice of medicine. CAT scans combine special x-ray equipment with sophisticated computers to produce images of the inside of the body. They are widely used, noninvasive medical tests that help physicians diagnose and treat numerous medical conditions. In 2000, the U.S. Food and Drug Administration (FDA) and the Conference of Radiation Control Program Directors (CRCPD) estimated that approximately 40 million CAT scans are performed annually.

In recent years, multiple articles have highlighted the increased risk of developing cancer from ionizing radiation. The risk increases with higher radiation doses, and accumulates with repeated scans. The 2007 American College of Radiology's white paper on radiation dose in medicine by Amis, et al., emphasizes the importance of addressing this issue, and proposes a plan to educate all stakeholders in the principles of radiation safety and appropriate utilization of imaging. In addition, in 2007 the Society for Pediatric Radiology joined forces with the American College of Radiology and several other medical societies to form the Alliance for Radiation Safety in Pediatric Imaging (the Image Gently Alliance). The charge of the Alliance is summarized in its mission statement: "…to raise awareness in the imaging community of the need to adjust radiation dose when imaging children."

Hospitals with computerized physician order entry systems (CPOE) have the unique opportunity to use decision support on radiation safety to influence a physician's ordering practice in real-time. CPOE and decision support technology have been successfully used to positively effect physician ordering behavior and improve patient safety in many aspects of patient care, including the ordering of radiology tests. An ideal decision support tool for radiation safety will educate the physician about the dangers of cumulative ionizing radiation, present the patient's image history, and guide the provider to the best modality that meets the patient's diagnostic needs with as little radiation exposure as possible. The design challenge is to create a decision support tool that appropriately protects our patients from overutilization of CAT scans, without inadvertently leading to underutilization of CAT scans or inappropriate utilization of alternative tests. This research protocol proposes to study one such design at a large, academic medical center.

ELIGIBILITY:
Inclusion Criteria:

* All inpatient providers who order a CAT Scan

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15969 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Ordering behavior in response to alert | After 6 months of data collection
  The proportion of patients that continue on with the CAT scan order, choose an alternative, or cancel the order in response to the radiation safety alert, as compared to control.

SECONDARY OUTCOMES:
Appropriateness of Imaging Test Ordered in Response to Safety Alert | After 6 months of data collection
  Decisions to proceed with the CAT scan order, choose an alternative or cancel the order will be evaluated for appropriateness by retrospective chart review by two independent radiologists. Discrepancies will be resolved by consensus.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Amis, MD, Principal Investigator — Montefiore Medical Center; Jason S Adelman, MD, MS, Study Director — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Amis ES Jr, Butler PF, Applegate KE, Birnbaum SB, Brateman LF, Hevezi JM, Mettler FA, Morin RL, Pentecost MJ, Smith GG, Strauss KJ, Zeman RK; American College of Radiology. American College of Radiology white paper on radiation dose in medicine. J Am Coll Radiol. 2007 May;4(5):272-84. doi: 10.1016/j.jacr.2007.03.002. PMID 17467608
- [Background] Goske MJ, Applegate KE, Bell C, Boylan J, Bulas D, Butler P, Callahan MJ, Coley BD, Farley S, Frush DP, McElveny C, Hernanz-Schulman M, Johnson ND, Kaste SC, Morrison G, Strauss KJ. Image Gently: providing practical educational tools and advocacy to accelerate radiation protection for children worldwide. Semin Ultrasound CT MR. 2010 Feb;31(1):57-63. doi: 10.1053/j.sult.2009.09.007. PMID 20102697